CLINICAL TRIAL: NCT05986500
Title: The GALAXY-1 Project: Galactose - the Ideal Carbohydrate Supplement for Exercise
Brief Title: The GALAXY-1 Project
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1-10-72-49-23
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2023-08

CONDITIONS: Healthy
Keywords: Galactose; Exercise; PET; Insulin
MeSH Terms: conditions — Motor Activity; Insulin Resistance | interventions — Galactose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Galactose (Experimental): The participants will receive a galactose infusion
  Interventions: Other: Galactose
- Saline (Experimental): The participants will receive a saline infusion
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Galactose — The participants will receive a galactose infusion (bolus: 6 mmol, infusion rate: 1 mmol/min)
  Arms: Galactose
Other: No intervention — The participants will receive a saline infusion
  Arms: Saline

SUMMARY:
"The understanding of the two sugars, glucose and fructose, has been thoroughly investigated regarding their impact on human metabolism during exercise. The consumption of the sugar galactose is an intriguing alternative and can be beneficial, especially for individuals with type 1 Diabetes, as it reduces the need for insulin to maintain normal blood sugar levels. Additionally, galactose oxidation rates during exercise are only 50-60% compared to glucose, primarily due to liver storage and/or the requirement for conversion to glucose in the liver before oxidation. This delay in metabolism can prevent hyperglycemia before exercise and provide extended protection against episodes of hypoglycemia during and after exercise through a moderate and prolonged glycemic response.

The purpose of this experiment is to investigate whether galactose is taken up by skeletal muscles and the heart in response to exercise or hyperinsulinemia. Using non-invasive 18F-FDGal PET, the investigators will examine this in a randomized controlled study design. The results could contribute to updating dietary recommendations, particularly for individuals with type 1 diabetes who struggle to maintain normal blood sugar levels during and after exercise."

DETAILED DESCRIPTION:
It is generally accepted that saccharides have to be converted into glucose before they can be oxidized and used to produce energy. As a result, non-glucose saccharides affect blood glucose levels differently than glucose. For example, the saccharide fructose requires hepatic conversion to glucose, causing more constant blood sugar levels and less risk of both glucose excursions and hypoglycemia during exercise. However, metabolization of fructose increases the risk of developing nonalcoholic fatty liver disease due to the stimulation of de novo lipogenesis and blocking of β-fatty acid oxidation. Consequently, a different carbohydrate source with the same glycemic profile as fructose but without the undesirable hepatic effects would be preferable. Galactose is the third of the three quantitively important dietary monosaccharides in a regular Western diet. Lactose (disaccharide of galactose and glucose) from dairy products is the primary source of dietary galactose, but galactose is also found in other food sources such as fruits and vegetables. While the impact of glucose and fructose on human metabolism has been extensively studied, there is limited knowledge of the effects of galactose as a nutritional supplement during or before exercise, and it is also unknown whether it can have clinical applications.

Intake of galactose or lactose instead of glucose prior to exercise may be advantageous, particularly for individuals with diabetes, since it lowers the insulin requirement to maintain euglycemia. Furthermore, galactose oxidation rates during exercise are only 50-60% compared to glucose, presumably due to hepatic storage and/or a requirement for conversion to glucose in the liver before oxidation. This delay in end-point metabolism could prevent hyperglycemia prior to exercise and at the same time provide prolonged protection from hypoglycemia during and after exercise via the prolonged and moderated glycemic response. In line with this, a recent study from the investigators' collaborator Gareth Wallis's group showed that lactose ingestion in relation to exercise increased fat oxidation and lowered carbohydrate oxidation compared to sucrose ingestion. Accordingly, ingestion of the lactose component - galactose - instead of regular glucose-containing carbohydrates is an intriguing option if blood glucose excursions are to be avoided. However, it is still unclear whether the beneficial metabolic effects of galactose are all caused by the hepatic delay in conversion to glucose or if galactose is also used directly by skeletal muscle as a source of energy. To address this, the investigators recently performed positron emission tomography (PET) pilot studies in two pigs using the galactose analogue 18F-FDGal to measure insulin-stimulated skeletal and cardiac muscle galactose uptake. Although muscle galactose uptake was clearly less than for glucose, it was evident that some uptake can be stimulated by insulin, particularly in the heart. These preliminary data question the current perception that galactose requires conversion to glucose in the liver before it can be utilized as a source of energy. However, studies in anesthetized pigs obviously cannot determine whether a similar direct muscle uptake of galactose can be stimulated by exercise per se, as is the case for glucose.

Purpose:

The purpose of this experiment is to investigate whether galactose is: 1) taken up by skeletal muscle and extra-hepatic organs, 2) if galactose uptake is affected by prior high intensity exercise with the purpose of depleting glycogen in the working skeletal muscle, and 3) if and to what extent insulin stimulates galactose uptake.

Methods:

Eight healthy participants will be studied twice in randomized order with 18F-FDGal PET scans during saline infusion (study day 1), and during a hyperinsulinemic-euglycemic clamp (study day 2). To stimulate galactose uptake in the femoral skeletal muscles, each participant will perform a 60-minute one-legged exercise prior to the PET scan. The non-exercised leg will serve as a control to quantify exercise-stimulated galactose uptake (Figure 2). During each study day, participants will receive a galactose infusion (bolus: 6 mmol, infusion rate: 1 mmol/min) to mimic concentrations of galactose similar to what can be achieved after galactose ingestion (1-2 mmol/L) (10). This design allows the investigators to quantify both the independent and combined effects of insulin and exercise on galactose uptake in skeletal muscle.

Volunteers:

Inclusion criteria:

1. Age 50-75 years
2. Males or post-menopausal females
3. BMI 18.5-30 kg/m2

Exclusion criteria:

1. Clinically significant heart, lung, kidney, liver, endocrine, or malignant disease based on information obtained during an initial screening visit as well as blood samples
2. Blood donation within the last 3 months
3. Smoking
4. Alcohol- or substance abuse
5. Participation in other clinical trials involving ionizing radiation within the last 6 months
6. Claustrophobia
7. Not being physically able to exercise one leg for one hour

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-75 years
2. Male or post-menopausal female
3. BMI 18.5-30 kg/m2

Exclusion Criteria:

1. Clinically significant heart, lung, kidney, kidney, liver, endocrine or malignant disease based on information obtained during an initial screening visit as well as blood samples
2. Blood donation within the last 3 months
3. Smoking
4. Alcohol- or substance abuse
5. Participation in other clinical trials involving ionizing radiation within the last 6 months
6. Claustrophobia
7. Not being physically able to exercise one leg for one hour

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Galactose uptake in skeletal muscle | Measurements will be made on each of the two study days
  Skeletal muscle galactose uptake rate (μmol/min/g) measured by 2-(18)F-fluoro-2-deoxy-d-galactose (18F-FDGal)

SECONDARY OUTCOMES:
Cardiac galactose uptake | Measurements will be made on each of the two study days
  Cardiac galactose uptake rate (μmol/min/g) measured by 2-(18)F-fluoro-2-deoxy-d-galactose (18F-FDGal)
Hepatic galactose uptake | Measurements will be made on each of the two study days
  Hepatic galactose uptake rate (μmol/min/g) measured by 2-(18)F-fluoro-2-deoxy-d-galactose (18F-FDGal)
Plasma glucose levels | Measurements will be made on a screening day and during each of the two study days
  Measured in blood samples
Skeletal muscle arterio-venous galactose balance | Measurements will be mader during each of the two study days
  Differences in arterio-venous galactose concentrations taken through catheters in both vv. famoralis and a. radialis

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus N, Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided